CLINICAL TRIAL: NCT04858048
Title: Use of the WALANT Anesthesia Technique for Forefoot Surgery.
Acronym: WALANT
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02531-38
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with general anesthesia performed during the forefoot surgery
  Interventions: Procedure: Anesthesia
- Group with WALANT anesthesia performed during the forefoot surgery
  Interventions: Procedure: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia — 2 types of anesthesia (general and WALANT) performed during the surgery

SUMMARY:
To compare the perioperative pain level with WALANT anesthesia versus general anesthesia during forefoot surgery.

DETAILED DESCRIPTION:
Orthopaedic foot and ankle surgery is typically performed while the patient is under general or regional anesthesia. The Wide Awake Local Anesthesia No Tourniquet (WALANT) technique is a local anesthesia technique used since 1980s in Canada for hand surgery. WALANT uses a combination of a local anesthetic and vasoconstrictor to induce anesthesia and hemostasis in the area of the surgical procedure in order to allow surgeries to be done without the use of tourniquet. This practice eliminates the need for the tourniquet due to the hemostatic effect of the vasoconstrictor. The administration of the local anesthetic is done as close as possible to the surgical site, which allows the mobility of the joint to be maintained, while having complete anesthesia. The retention of mobility and the absence of a tourniquet improve patient comfort.

The main objective of this prospective study is to evaluate the perioperative pain level with WALANT anesthesia compared to general anesthesia during forefoot surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient with scheduled forefoot surgery

Exclusion Criteria:

* Protected patient : major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scheduled forefoot surgery.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Perioperative
  Measure of the pain using the VAS pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: François LAVIGNE, Principal Investigator — Hôpital Privé Saint Martin
Locations (1):
- Hôpital Privé saint Martin, Caen, France

IPD SHARING:
Plan to Share IPD: No